CLINICAL TRIAL: NCT07112287
Title: MyeloGen: Germline Testing for Predisposition to Myeloid Malignancies
Brief Title: Germline Testing for Predisposition to Myeloid Malignancies
Acronym: MyeloGen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Reilly (Other)
Collaborators: Broad Institute of MIT and Harvard (Other)
Responsible Party: Sponsor-Investigator, Christopher Reilly, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-218
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Myeloid Malignancy; Genetic Predisposition to Disease; Myeloid Hematological Malignancies
Keywords: Myeloid Malignancies; Genetic Predisposition to Disease
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- MyeloGen Germline Testing Group (Experimental): Enrolled participants will complete:
  * Baseline visit with questionnaires, educational video, and punch skin biopsy
  * Negative genetic test results notification via mail
  * Positive genetic results will be followed up by an appointment with a genetic counselor or physician
  * Post-results questionnaires
  * Follow up via medical records for up to 2 years from time of study consent.
  Interventions: Device: MyeloGen Gene Panel

INTERVENTIONS:
Device: MyeloGen Gene Panel — The MyeloGen Gene Panel is investigational Germline genetic testing using skin fibroblasts.
  Other Names: Custom hereditary cancer gene panel

SUMMARY:
The goal of this research study is to evaluate the feasibility of germline genetic testing using the investigational MyeloGen Gene Panel in adult participants diagnosed with myeloid malignancies.

DETAILED DESCRIPTION:
This prospective, single arm study aims to evaluate the feasibility of germline genetic testing using the investigational MyeloGen Gene Panel in adult participants diagnosed with myeloid malignancies. Investigators hope to learn how to best incorporate routine genetic testing in clinical care for participants with blood cancers, regardless of personal or family history of blood cancer.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, and punch skin biopsies.

It is expected that about 200 people will take part in this research study.

The laboratory sponsor of this protocol is Broad Clinical Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Participants must have histologically confirmed myeloid malignancy OR bone marrow failure within the last 6 months prior to screening.
* Ability to understand and provide a signed and completed consent document in English.

Exclusion Criteria:

* Participants who cannot safely undergo clinically indicated skin biopsy as adjudicated by the study team.
* Participants who have previously undergone germline genetic testing for predisposition to myeloid malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
Successful Completion Rate | Up to 10 weeks
  Successful completion rate of germline genetic testing will be defined as the proportion of participants who return genetic test results within 10 weeks of study consent, which would require there be no excessive delays in obtaining a skin biopsy.

SECONDARY OUTCOMES:
Number of Participants with Positive Results | Up to 12 weeks
  A "positive" result indicating a pathogenic or likely pathogenic variant was detected. This will also include Variants of Unknown Significance (VUSs) with supporting pathogenic criteria per American College of Medical Genetics guidelines (ACMG).
Patient Reported Outcome of Germline Genetic Testing based on GST Survey | Up to 60 days
  Participants will complete the GST survey 1 (after the educational video and skin biopsy) and GST survey 2 between 45-60 days after disclosure of genetic test results. GST survey answers will be converted to a 5-point scale: 1- Disagree strongly, 2-Disagree, 3-Neither Agree or Disagree, 4-Agree, 5- Agree strongly.
Number of Participants with an Identified Germline Predisposition on Generic Testing Who Haven't Met NCNN Guideline-based Germline Genetic Testing Recommendations | Up to 12 weeks
  NCCN guideline-based eligibility for germline genetic testing will be assessed using the following criteria and manual review of participants' medical record, 1) Participants with Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) less than age 50, 2) Hypoplastic MDS regardless of age; 3) History of aplastic anemia, 4) Documented suspicion of a possible germline predisposition to myeloid malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Reilly, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu